CLINICAL TRIAL: NCT06074809
Title: Clinical Trial on the Treatment of Menopausal Syndrome With Chinese Medicine Gui-zhi-fu-ling-wan With Variation and the Mechanism of Anti-inflammation and Body Surface Temperature Distribution
Brief Title: RCT on the Treatment of Menopausal Syndrome With Chinese Medicine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zhang Hongwei, School of Chinese Medicine, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Menopause study
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Menopause
Keywords: Traditional Chinese medicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese medicine treatment group (Experimental): Chinese medicine will be administered to patients in this group.
  Interventions: Drug: Modified Guizhi Fuling granules
- Placebo group (Placebo Comparator): Placebo will be administered to patients in this group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Modified Guizhi Fuling granules — Modified Guizhi Fuling granules will be orally administered to patients in the TCM treatment group twice a day throughout the treatment period, which lasts for 8 weeks.
  Other Names: Chinese medicine
  Arms: Traditional Chinese medicine treatment group
Other: Placebo — Placebo will be orally administered to patients in the placebo group twice a day throughout the treatment period, which lasts for 8 weeks.
  Arms: Placebo group

SUMMARY:
This is a double-blinded, randomized, placebo-controlled clinical trial. Subjects will be randomly assigned to the treatment group (Modified Guizhi Fuling granules) or placebo group (Placebo granules) for 8 weeks. Outcomes will be measured at week 8 and week 12.

DETAILED DESCRIPTION:
Menopausal syndrome is a series of symptoms caused by ovarian follicles degeneration that occurs before or after menopause. These symptoms include central nervous system-related disorders (such as hot flashes, insomnia, depression, anxiety, etc.); metabolic, weight, cardiovascular and musculoskeletal changes; urogenital and skin atrophy; and sexual dysfunction.

Some previous studies have investigated the possibilities of using traditional Chinese medicine (TCM) for the treatment of menopausal syndrome. However, due to the limitations of previous clinical research, more evidence is required to support the efficacy of TCM treatment. Therefore, we propose to conduct a randomized, double-blinded, placebo-controlled clinical trial here, with the hope of objectively assessing the efficacy and safety of using TCM to treat menopausal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with age between 40 and 60 years old;
* For those who have symptoms of primary menopause (irregular menstruation lasting for more than 6 months, or absence of menstrual periods for more than 3 months)
* The score of the physical symptoms in Greene Climacteric Symptom Score (GCS) is 6 or above (average level);
* Have moderate level (affecting certain level of daily activity) or severe (cannot carry out daily activity) hot flashes, defined as transient sensations of heat, sweating, flushing, anxiety and chills lasting for 1-5 minutes;
* Diagnosed Deficiency of Kidney essence and static blood in Lower Jiao by Chinese medicine practitioner
* Agreed to receive Chinese medication or placebo for 2 months upon randomization.

Exclusion Criteria:

* The menopausal syndrome caused by surgical operations or medications (such as chemotherapy, gonadotropin-releasing hormone agonists, etc.).
* Have received estrogen treatment in the past 2 months;
* Have received any medication for treating menopause in the past month, including herbs, non-prescribed drugs, supplements, or change of diet to consume more legumes;
* Known serious emotional, mental or psychological disorders that may affect the study;
* During pregnancy, pre-pregnancy period, or lactation period;
* Known history of allergy to any traditional Chinese medicine;
* Have received anticoagulant or antiplatelet drugs in the past month;
* Known history of some certain serious medical disease, such as cardiovascular disease, liver or renal dysfunction, diabetes, cerebrovascular disease, blood disorders, with unstable conditions;
* Chinese medicine pattern combined with damp phlegm or damp heat, or only deficiency of Yin blood or absence of static blood pattern.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Greene Climacteric Scale (Chinese version) | Week 8
  Greene Climacteric Scale (GCS) is one of the most common scales used to assess menopause. It includes four aspects of symptoms: vasomotor, somatic, psychological, and sexual response. This scale consists of 21 symptoms that can be assessed by patients themselves. The scoring from 0 to 3 in each item, indicates 'Not at all', 'A little bit', 'Much', and 'Very much' respectively.

SECONDARY OUTCOMES:
Short-Form Health Survey, SF-12v2 (Chinese version) | Week 8
  The SF-12v2 is the brief version of SF-36, consisting of 12 questions related to our physical, mental health and functionality. It is used as a supportive tool to comprehensively assess the health status of the patient. Scores range from 0 to 100, with higher scores representing better self-reported health.
Short-Form Health Survey, SF-12v2 (Chinese version) | Week 12
  The SF-12v2 is the brief version of SF-36, consisting of 12 questions related to our physical, mental health and functionality. It is used as a supportive tool to comprehensively assess the health status of the patient. Scores range from 0 to 100, with higher scores representing better self-reported health.
Temperature change of face, limbs and abdomen | Week 8
  The peripheral temperature of the face, limbs and abdomen of the patients will be measured by a thermographic camera.
Temperature change of face, limbs and abdomen | Week 12
  The peripheral temperature of the face, limbs and abdomen of the patients will be measured by a thermographic camera.
Level change of sex hormones | Week 8
  Level change of Estradiol (E2) and Follicle-stimulating hormone (FSH) will be measured between baseline and week 8.
Level change of sex hormones | Week 12
  Level change of Estradiol (E2) and Follicle-stimulating hormone (FSH) will be measured between baseline and week 12.
Level change of inflammatory markers | Week 8
  Level change of the serum inflammatory factors: high-sensitivity C-reactive protein (hsCRP), Interleukin 6 (IL-6) , Interleukin 8 (IL-8) and Tumor necrosis factor-α (TNF-α) will be measured from baseline to week 8.
Level change of inflammatory markers | Week 12
  Level change of the serum inflammatory factors: high-sensitivity C-reactive protein (hsCRP), Interleukin 6 (IL-6) , Interleukin 8 (IL-8) and Tumor necrosis factor-α (TNF-α) will be measured from baseline to week 12.
Greene Climacteric Scale (Chinese version) | Week 12
  Greene Climacteric Scale (GCS) is one of the most common scales used to assess menopause. It includes four aspects of symptoms: vasomotor, somatic, psychological, and sexual response. This scale consists of 21 symptoms that can be assessed by patients themselves. The scoring from 0 to 3 in each item, indicates 'Not at all', 'A little bit', 'Much', and 'Very much' respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhang, PhD, Principal Investigator — School of Chinese Medicine
Locations (1):
- School of Chinese Medicine, Shatin, Hong Kong